CLINICAL TRIAL: NCT02897102
Title: Effects of a Training Program Based on Abacus and Other Activities in Healthy Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Rogerio Panizzutti, Professor, Universidade Federal do Rio de Janeiro
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 257651
Record Dates: First submitted 2016-08-18; First posted 2016-09-13 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Active Comparator): The individuals in the control group chose to participate in different group activities: ballroom dancing (5 participants), belly dancing (4 participants), chorus (16 participants), Spanish classes (8 participants) and chorus and Spanish classes (6 participants). The activities were offered once per week in 2 hours classes for 35 weeks and were held between April and November of 2013.
  Interventions: Other: Different group activities
- Training group (Experimental): was offered in one weekly class for 2 hours for 35 weeks between April and November of 2013. The first 50 minutes were spent performing exercises with the abacus, with increasing difficulty. One or two of the following activities followed the abacus training: playing games, neurobic and group dynamics.
  Interventions: Behavioral: Training

INTERVENTIONS:
Behavioral: Training — Training program based on abacus and other activities
  Arms: Training group
Other: Different group activities — ballroom dancing (5 participants), belly dancing (4 participants), chorus (16 participants), Spanish classes (8 participants) and chorus and Spanish classes (6 participants).
  Arms: Control group

SUMMARY:
The aim of this study was to investigate the effects of a structured program, which was based on abacus training associated with other activities, administered as weekly group classes over a 7 month period in older adults.

DETAILED DESCRIPTION:
Cognitive stimulating activities are often recommended for older adults; however, little is known regarding the effects of these activities on cognition, motivation and quality of life in this population. The aim of this study was to investigate the effects of a structured program, which was based on abacus training associated with other activities, administered as weekly group classes over a 7 month period in older adults. Eighty-eight older adults were enrolled in an open-label controlled clinical trial to evaluate the effects of this training program on cognition, motivation and quality of life. Training had a significant effect over time; the training group maintained their level of performance on verbal learning and memory tasks, whereas the control group exhibited a significant decrease in performance from baseline to post-intervention. The subjects in the training group were more motivated to learn at study entry; however, the training had no significant effect on motivation or quality of life. Abacus training associated with other activities may benefit verbal learning and memory in older adults. Additional studies with longer follow-ups are necessary to determine whether the results of this training will have a positive effect on the lives of older adults.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* Score ≥ 26 on the Mini-Mental State Examination
* Portuguese as a native language.

Exclusion Criteria:

* A neurological or serious medical condition that would prevent participation in the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2013-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Reasoning score change | After 7 month
  Reasoning score change will be measured using the Z-score of Matrix Reasoning subtest of the BETA III
Attention score change | After 7 month
  Attention score change will be measured using the average of the Z-scores of the Codes subtest of the BETA III and the Cogstate Identification Task
Speed of processing score change | After 7 month
  Speed of processing score change will be measured using the Z-score of the Cogstate Detection Task
Working memory score change | After 7 month
  Working memory score change will be measured using the average of the Z-scores of the Cogstate One Back and Two Back tasks
Verbal learning and memory score change | After 7 month
  Verbal learning and memory score change will be measured using the average of the Z-scores of the Cogstate International Shopping List and International Shopping List - Delayed Recall tasks
Visual learning and memory score change | After 7 month
  Visual learning and memory score change will be measured using the average of the Z-scores of the Cogstate Continuous Paired Associate Learning, One Card Learning and Groton Maze Learning Test - Delayed Recall tasks
Executive function score change | After 7 month
  Executive function score change will be measured using the average of the Z-scores of the Cogstate Groton Maze Learning Test and Set Shifting Task

SECONDARY OUTCOMES:
Motivation | After 7 months
  Evaluated using the self-concept scales of cognitive competence and self-learning
Quality of life | After 7 months
  Evaluated using the control, autonomy, self-realization, and pleasure scale (CASP-19)

IPD SHARING:
Plan to Share IPD: No